CLINICAL TRIAL: NCT03386201
Title: FLuorescence Cholangiography Using Methylene Blue
Acronym: FLoCaMB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, DrThomasBarnes, Clinical Research Fellow, University of Oxford
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13174
Record Dates: First submitted 2017-12-18; First posted 2017-12-29 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Bile Duct Injury
Keywords: Laparoscopic cholecystectomy; Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravenous methylene blue (Experimental)
  Interventions: Drug: Intravenous Methylene blue

INTERVENTIONS:
Drug: Intravenous Methylene blue — Methylene blue fluorescence cholangiography during laparoscopic cholecystectomy

SUMMARY:
Open label prospective, non-randomised proof of principle study assessing the use of methylene blue fluorescence cholangiography.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Undergoing laparoscopic cholecystectomy

Exclusion Criteria:

* Patient who is unable or unwilling to give informed consent
* Known allergy to methylene blue
* Risk of serotonin syndrome (taking SSRI / G6PD deficiency / previous serotonin syndrome)
* Significant renal failure
* Pregnant / planning pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Concordance of surgeon anatomy definition with fluorescence outline | Intraoperative (At end of laparoscopic cholecystectomy)

SECONDARY OUTCOMES:
Signal to background ratio over time throughout laparoscopic cholecystectomy | 0, 10, 20, 30, 40, 50, 60, minutes and at 10 minute intervals thereafter post injection of methylene blue

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No